CLINICAL TRIAL: NCT04383600
Title: Efficacy of Micro-osteoperforations on the Rate of Maxillary Canine Retraction: A Randomized Controlled Trial
Brief Title: Flapless Mops for Acceleration of Canine Retraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Akram Elawady (Other)
Responsible Party: Sponsor-Investigator, Ahmed Akram Elawady, Principal Investigator, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100
Record Dates: First submitted 2020-05-02; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Dental Malocclusions; Angle Class II, Division 1; Bimaxillary Protrusion
Keywords: MOPs; micro-osteoperforation; acceleration; orthodontic tooth movement
MeSH Terms: conditions — Malocclusion, Angle Class II | interventions — morpholinopropane sulfonic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional side (No Intervention): Canine retraction was commenced without micro-osteoperforations.
- Mops side (Experimental): Canine retraction was commenced with micro-osteoperforations.
  Interventions: Procedure: Micro-osteoperforation

INTERVENTIONS:
Procedure: Micro-osteoperforation — three flapless micro-osteoperforations was performed distal to the maxillary canine before starting retraction.
  Other Names: Mops
  Arms: Mops side

SUMMARY:
The aim of the present clinical study was directed to evaluate the effectiveness of micro-osteoperforations on the rate of canine retraction; in addition, the potential risk for root resorption during maxillary canine retraction.

DETAILED DESCRIPTION:
The aim of the present clinical study was directed to evaluate the effectiveness of micro-osteoperforations on the rate of canine retraction; in addition, the potential risk for root resorption during maxillary canine retraction.

This study was conducted on a total sample of 24 canines of 12 patients, 8 females and 4 males, with mean age was 16.17 ± 2.29 years old who required therapeutic extraction of maxillary 1st premolars and canine retraction. They were selected randomly from the Outpatient Clinic, Department of Orthodontics, Faculty of Dental Medicine (Boys), Al-Azhar University, Cairo, Egypt.

Both maxillary canines, in each patient, were randomly assigned to either an experimental side or the control side in a simple split-mouth design. In the experimental side, micro-osteoperforations was performed distal to the maxillary canine before starting retraction, while the canines in the contralateral control side were retracted without micro-osteoperforations.

Extraction was done at the start of the treatment, and before fitting of the orthodontic appliance. Then upper dental arches were leveled and aligned using conventional sequences of wires.

Three flapless micro-osteoperforations was performed by using orthodontic miniscrews distal to the maxillary canines in the experimental side before starting retraction. Each perforation was 1.6 mm in diameter and 3-4 mm depth into the bone. Canines were completely retracted on 0.016 × 0.022 ̋ stainless steel wires by using closed coil spring delivered 150 gm force.

Patients were followed up every 28 days until complete canine retraction. Routine orthodontic records were obtained for each patient before treatment.

Additionally, a full skull CBCT images were taken before treatment and immediately after canine retraction.

The rate of canine retraction was assessed clinically; in addition, cone beam CT (CBCT) scans were used to assess the amount of canine retraction root length changes. Also anchorage loss of first permanent molars were assessed.

The treatment results were compared clinically and radiographically (CBCT).

ELIGIBILITY:
Inclusion Criteria:

1. An age ranged between 14 to 18 years.
2. Class II division 1 malocclusion or Class I bimaxillary protrusion with mild or no crowding. Wherever crowding was present, it was symmetrical on both sides of the arch.
3. Patients who diagnosed to require extraction of at least maxillary first premolars bilaterally as a part of their treatment plan.
4. Complete permanent dentition (3rdmolars were not included).
5. Good oral and general health.
6. No history of periodontal problems.
7. No therapeutic intervention planned involving intermaxillary or other intraoral or extraoral appliances during the study period.

Exclusion Criteria:

1. Blocked out or impacted maxillary canines.
2. Transverse and/or vertical skeletal dysplasia or craniofacial anomalies.
3. Systemic diseases or regular use of medications that could interfere with orthodontic treatment.
4. Previous orthodontic treatment.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-06-05 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | change from start of canine retraction until complete space closure up to 6 months
  Clinically, patients were evaluated immediately before canine retraction and every 4 weeks till complete space closure (complete canine retraction).
  It was based on measuring the distance between the contact points on the distal surface of the canines and the contact points on mesial surface of the second premolars.
Canine root length changes | change from start of orthodontic treatment until complete space closure up to 9 months
  The CBCT scans were taken before orthodontic treatment and after complete space closure (canine retraction) to be analyzed for assessment of Canine root length changes.
  The root length was measured along the axis of the root, perpendicular to a line connecting the buccal and palatal cemento-enamel junction CEJ in sagittal view

SECONDARY OUTCOMES:
Anchorage loss of maxillary first permanent molars. | change from start of orthodontic treatment until complete space closure up to 9 months
  mesial movement of maxillary first permanent molars bilaterally was measured before orthodontic treatment and after complete space closure ( canine retraction) on CBCT scan which were taken before orthodontic treatment and after complete canine retraction The distance measured along perpendicular from distal surface of 1st permanent molar to Ptv plane

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El Awady, Principal Investigator — Al-Azhar University
Locations (1):
- Al azhar university, Cairo, Egypt